CLINICAL TRIAL: NCT04897802
Title: Identification and Clinical Relevance of an Oxytocin Deficient State: a Randomized, Crossover, Placebo-controlled, Proof-of-concept, Physiopathological Study (GLP1 Study)
Brief Title: Identification and Clinical Relevance of an Oxytocin Deficient State (GLP1 Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIBSP-OXI-2020-102
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-03

CONDITIONS: Hypopituitarism; Central Diabetes Insipidus; Panhypopituitarism; Psychological Disorder; Social Isolation; Hypothalamic Diseases; Pituitary Diseases; Oxytocin Deficiency
Keywords: oxytocin; hypopituitarism; diabetes insipidus; hypothalamic-pituitary diseases; psychopathology; exenatide
MeSH Terms: conditions — Hypopituitarism; Diabetes Insipidus, Neurogenic; Combined Pituitary Hormone Deficiency; Mental Disorders; Social Isolation; Hypothalamic Diseases; Pituitary Diseases; Diabetes Insipidus | interventions — Exenatide; Organization and Administration; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: GLP1-RA administration (Experimental): A single dose of 10 mcg of GLP1-RA (exenatide) will be injected subcutaneously and samples will be collected over 2 hours (15 (T15), 30 (T30), 45 (T45), 60 (T60'), 90 (T90) and 120 (T120) minutes) after GLP1-RA:placebo administration to assess OT secretory patterns
  Interventions: Drug: Experimental: GLP1-RA (exenatide) administration
- Control: Placebo administration (Placebo Comparator): Sodium Chloride 0.9% will be administered subcutaneously at equivalent volume than GLP1-RA (exenatide) administration
  Interventions: Drug: Control: Placebo administration

INTERVENTIONS:
Drug: Experimental: GLP1-RA (exenatide) administration — a single dose of 10 mcg of GLP-RA (exenatide) will be administered subcutaneously and samples to assess OT secretory patterns will be collected over 2 hours
  Other Names: exenatide administration
  Arms: Experimental: GLP1-RA administration
Drug: Control: Placebo administration — Sodium Chloride 0.9% will be administered subcutaneously at equivalent volume than 10 mcg of exenatide
  Other Names: placebo administration (sodium chloride)
  Arms: Control: Placebo administration

SUMMARY:
Oxytocin (OT) is a hypothalamic peptide that enters the peripheral circulation via the posterior pituitary gland. OT plays a key role in regulating appetite, psychopathology, prosocial behavior and sexual function. Hypopituitarism is associated with increased obesity, increased psychopathology, sexual and prosocial dysfunction despite appropriate hormone replacement. A few studies suggest the existence of a possible OT deficient state in hypopituitarism. In animal models, glucagon-like peptide 1 (GLP1) has shown to increase OT release.

This study is designed to evaluate OT values after administration of GLP1 in adults (healthy volunteers and patients with hypopituitarism).

The investigators hypothesize that OT response will be blunted following GLP1 receptor agonist (GLP1-RA) in patients with hypopituitarism compared to healthy controls.

DETAILED DESCRIPTION:
This research is focused on two groups of participants: healthy controls (HC) and hypopituitary patients (HYPO) with at least one symptom of hypothalamic damage, presumably at highest risk for OT deficiency.

The aim is to improve knowledge on the physiology and patho-physiology of endogenous OT secretion in hypopituitary patients compared to healthy controls using a randomized, single-blind, crossover assignment (GLP1-RA vs placebo), placebo-control design.

Clinical implications of secretory OT dynamics and release under different stimuli using validated questionnaires to evaluate psychopathology, socio-emotional functioning, disordered eating behavior, impaired quality of life and sexual dysfunction, will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypopituitarism (HYPO) (>1 pituitary hormone deficiency) and stable hormone replacement for the prior three months
* At least one clinical sign of hypothalamic damage
* Female participants will be done in the early to midfollicular phase

Exclusion Criteria:

* uncorrected hormone deficiency
* creatinine >1.5mg/dL
* alanine aminotransferase (ALT) or aspartate amino transferase (AST) >2.5x upper limit of normal
* hematocrit less than 30%
* suicidality or active psychosis
* participation in a trial with investigational drugs within 30 days
* using a high glucocorticoid dose
* Any type of diabetes mellitus
* Obese patients on GLP1-RA therapies
* vigorous physical exercise
* alcohol intake within 24 hours before the study participation
* evidence of any acute illness or any illness that the Investigator determines could interfere with study participation or safety
* pregnancy or breastfeeding for last 8 weeks
* known allergies towards GLP1-RA
* patients refusing or unable to give written informed consent
* Additionally for healthy controls: the presence of brain or pituitary tumor, radiation involving the hypothalamus or pituitary, history of hypopituitarism or receiving testosterone or glucocorticoids esters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in oxytocin concentration (pg/mL) | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in oxytocin concentration (pg/mL) after administration of 10 µg of GLP1-RA (exenatide) or 0.9% sodium chloride (NaCl)

SECONDARY OUTCOMES:
Maximal change in oxytocin concentration (pg/mL) | Within the two hours after the injection
  Change in oxytocin concentration (pg/mL) after administration of 10 µg of GLP1-RA (exenatide) or 0.9% NaCl
Overall oxytocin secretion (pg/mL) | Within the two hours after the injection
  Oxytocin area under the curve after administration of 10 µg of GLP1-RA (exenatide) or 0.9% NaCl
Change in glucose concentration (mg/dL) | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in glucose concentration (mg/dL) after administration of 10 µg of GLP1-RA (exenatide) or 0.9% NaCl
Change in insulin concentration (pmol/L) | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in insulin concentration (pmol/L) after administration of 10 µg of GLP1-RA (exenatide) or 0.9% NaCl
Mood assessment | Baseline
  Association between Beck Depression Inventory-2 score (range from 0 to 63, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)
Quality of life assessment | Baseline
  Association between 36-item Short Form Health Survey score (range from 0 to 100, the higher scores indicate better health status) and baseline oxytocin concentration (pg/mL)
Impulsivity assessment | Baseline
  Association between Barratt Impulsiveness Scale (range from 30 to 120, higher scores indicate greater impulsivity) and baseline oxytocin concentration (pg/mL)
Alexithymia assessment | Baseline
  Association between Toronto Alexithymia scales-20 score (range from 20 to 100, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Aulinas, MD PhD, Principal Investigator — IR-Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain